CLINICAL TRIAL: NCT03393130
Title: Perioperative Research Into Memory GENomics in the Intensive Therapy Unit: Alzheimer's (PRIMoGenITA): The Genomics of Cognitive Impairment After Admission to a Burns Intensive Care Unit
Brief Title: Perioperative Research Into Memory, Genomics in the Intensive Therapy Unit: Alzheimer's
Acronym: PRIMoGenITA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Marcela P. Vizcaychipi, Principle Investigator, Chelsea and Westminster NHS Foundation Trust
Other Study IDs: C&W17/059
Record Dates: First submitted 2017-12-11; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Cognitive Impairment; Apolipoprotein E, Deficiency or Defect of; Critical Illness; Burns; Young Adult
Keywords: Burns; Young Adult; Cognitive Impairment; Apolipoprotein E, Deficiency or Defect of; Intensive Care Neurological Disorder; Quality of Life; Inflammation, Brain
MeSH Terms: conditions — Cognitive Dysfunction; Apolipoprotein E, Deficiency or Defect of; Critical Illness; Burns; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants possessing APOE-ε4: Young adults who have suffered a severe burn injury necessitating intensive care admission 5 to 10 years previously, who possess at least one copy of the APOE-ε4 allele.
  Interventions: Diagnostic Test: APOE genotyping
- Participants not possessing APOE-ε4: Young adults who have suffered a severe burn injury necessitating intensive care admission 5 to 10 years previously, who do not possess a copy of the APOE-ε4 allele.
  Interventions: Diagnostic Test: APOE genotyping

INTERVENTIONS:
Diagnostic Test: APOE genotyping — APOE genotyping and broad cognitive assessment expressed as a median T-score of the following tests (with cognitive domains assessed in brackets) Trail Making Part A (processing speed), Trail Making Part B (executive function), One Back test (working memory), List Learning Task (Immediate recall, visual learning, delayed recall and recognition discrimination).
  Other Names: Neurocognitive testing

SUMMARY:
The current central dogma of long-term cognitive impairment after intensive care admission suggests an underlying neuroinflammatory dysregulation affecting neuronal function. This pathological process has not been fully elucidated and there has been little research into its genetic associations.

Alzheimer's disease (AD) causes cognitive impairment through a process of abnormal beta amyloid deposition and neuronal death through localised activation of the innate immune system. It is the most prevalent disease affecting cognition. The Apolipoprotein E (APOE) gene is implicated in the progression of late-onset Alzheimer's disease and is a recognised neuroinflammatory modulator. It is possible that young individuals exposed to high levels of inflammation may experience an acceleration of this process. This study sets out to look for an association between APOE-∈4 possession and poor cognitive outcome after a major burn injury and intensive care admission.

DETAILED DESCRIPTION:
Long-lasting post-operative cognitive dysfunction (POCD) is now a well-recognised complication of surgery, anaesthesia and critical care. It has been shown that cognitive impairment in critical care survivors can be worse than cohorts diagnosed with Mild Cognitive Impairment and approaching those suffered moderate Traumatic Brain Injury. POCD most significantly impacts upon the elderly, comorbid and those with pre-existing cognitive impairment, and has a socially and psychologically significant impact on quality of life.

The current central dogma suggests an underlying neuroinflammatory dysregulation affecting neuronal function. However, the underlying pathological processes have not yet been fully elucidated. Although some risk factors have been recognised we cannot accurately predict outcome, suggesting other unidentified determinants. The discovery of further risk factors would allow new insights into the underlying mechanism, and open up future avenues of investigation and potential interventions.

Thus far, little work has been performed looking into the impact of genomics on cognitive outcome after critical care. There are an estimated 20,000 protein coding genes in the human genome. Such large numbers of whole exome sequence variables necessitate using either an extremely large population or testing a small number of candidate genes. Critical Care research is hampered by small population sizes, ruling out whole genome analysis. The ideal candidate gene would be a known modulator of neuroinflammation, synthesised in the central nervous system (or able to traverse the blood-brain barrier) and have a known association with cognitive impairment. In terms of feasibility it should have relatively high incidence allele proportions, and be modifiable for in order to test any association for causality.

The most common gene associated with cognitive impairment is APOE, which codes for apolipoprotein E (ApoE). There are three common alleles of the APOE gene: APOE-∈2, APOE-∈3 and APOE-∈4. Possession of an APOE-∈4 allele increases the risk of developing late-onset Alzheimer's Disease. ApoE demonstrates immunomodulatory properties both systemically and in the central nervous system. It is secreted by astrocytes and oligodendrocytes after brain injury and is implicated in the cholesterol distribution necessary for membrane growth after axonal injury. ApoE-deficient murine glial cultures express more nitric oxide (NO) and Tissue Necrosis Factor α (TNFα) after simulated injury (LPS / closed head injury) than wild-type cells. Incubating the deficient glial cultures in recombinant apoE suppresses the TNF-α expression. This suppression occurred to a much greater extent with recombinant apoE-∈3 and apoE-∈2 than with apoE-∈4. Finally, microglia treated with secreted amyloid precursor protein α (sAPP-α, a secreted derivative of β amyloid precursor protein (β-APP)) will produce higher levels of activation markers and enhance the production of neurotoxins. This effect can be blocked by prior incubation apoE3, but not with apoE4. Administration of peripheral ApoE mimetic peptide (a truncated protein able to traverse the blood brain barrier) suppresses systemic and brain Il-6 and TNFα levels. Lastly, ApoE isoforms also have different affects on cholinergic neuron destruction, through increased synthesis and reduced elimination of amyloid beta.

Critical care patients typically experience systemic inflammation secondary to sepsis, surgery or trauma, or a combination of the three. Central nervous system (CNS) ApoE mRNA expression is upregulated in wild-type mice exposed to repeated restraint stress. As such, it is possible that APOE genotype may influence cognitive outcome through mediation of the neuroinflammatory response. The APOE-∈4 allele is known to increase the risk of POD after surgery and to increase the duration of delirium in the intensive care unit (ITU). The presence and duration of post-operative delirium (POD) are recognised predictors of long-term cognitive impairment (LTCI). Neither the incidence of delirium nor LTCI according to APOE genotype have been investigated in critical care patients.

More recently, burns intensive care (BICU) survivors have also been shown to develop LTCI following discharge with an associated reduction in quality of life.

The incidence of cognitive impairment amongst severe burns patients is comparable to ARDS cohorts, but in a younger and less comorbid group. Patients with severe burns develop large magnitude systemic inflammatory reactions secondary to their injury. This is perpetuated by multiple surgeries and a high incidence of nosocomial infections. This cohort provides a unique group of relatively young individuals with comparable injuries and minimal pre-morbid comorbidity or cognitive impairment. As such, they represent a less varied population than general adult ITUs. It is also unusual to find evidence of AD, vascular dementia or Parkinson's dementia in younger age brackets. This reduces the confounding factors that typically impede critical care clinical research and any association between APOE-∈4 and ITU LTCI may therefore infer a common pathological process.

We hypothesise that severe burn patients who possess an APOE ε4 allele are more susceptible to long term cognitive impairment following their injuries, and that this will impact significantly on their quality of life.

With this study we aim to: assess neurocognitive function following a severe burn; more specifically processing speed, executive function, working memory, immediate recall and delayed recall; assess our sample population APOE genotype; and investigate the association between APOE genotype and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Consenting individual
* Burn injury >15% total body surface area
* Admission to a Burns Intensive Care Unit between Jan 2007- Jan 2012
* Intubated and ventilated during the admission

Exclusion Criteria:

* Patients admitted to BICU with Toxic Epidermal Necrolysis Syndrome or Steven-Johnson Syndrome
* Head trauma
* Currently held under the 2007 Mental Health Act (UK) or Section 5150 of the California Welfare and Institutions Code (USA).
* Currently receiving formal psychiatric treatment (including involvement in a Personality Disorder Unit, being under voluntary section, current re-occurrence of chronic self-harm)
* Current imprisonment
* Current substance abuse (within two weeks of assessment)
* Patients unable to understand plain verbal and written English.

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Consenting young adults who suffered a severe burn injury necessitating intensive care admission 5-10 years previously.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
APOE genotype | Twelve month recruitment window
  Possession of an APOE-ε4 allele

SECONDARY OUTCOMES:
Cognitive impairment | Twelve month recruitment window
  Above or below the median cognitive score
Short Form of the Informant Questionnaire on Cognitive Decline in the Elderly score | Twelve month
  Estimate of premorbid cognitive function (confounder)
Adapted American Psychiatric Association National Institute on Drug Abuse Modified Alcohol, Smoking and Substance Involvement Screening Test (APA NM-ASSIST) | Twelve month
  Substance misuse index
Health Utilities Index 3 (HUI-3) score | Twelve month
  Quality of life index
Patient Health Questionnaire 9 (PHQ-9) score | Twelve month
  Depression index
Generalised Anxiety Disorder 7 (GAD 7) score | Twelve month
  Anxiety index
Trauma Screening Questionnaire (TSQ) score | Twelve month
  Post-traumatic stress index

CONTACTS AND LOCATIONS:
Overall Officials: Marcela P Vizcaychipi, MD PhD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided